CLINICAL TRIAL: NCT05533528
Title: Periodontal Granulation Tissue Preservation in Surgical Periodontal Disease Treatment. a Randomized Clinical Trial
Brief Title: Periodontal Granulation Tissue Preservation in Surgical Periodontitis Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Antonio José Ortiz Ruiz, MD, Professor and researcher, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3111/2020
Record Dates: First submitted 2022-09-05; First posted 2022-09-09 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-12

CONDITIONS: Periodontal Pocket; Periodontal Diseases; Periodontal Bone Loss
MeSH Terms: conditions — Periodontal Pocket; Periodontal Diseases; Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Access flap periodontal surgery
  Interventions: Procedure: periodontal surgery
- Test (Experimental): Access flap periodontal surgery and periodontal granulation tissue debridement.
  Interventions: Procedure: periodontal surgery

INTERVENTIONS:
Procedure: periodontal surgery — A sulcular incision will be made in the affected teeth, followed by an incision from the buccal aspect in the mid-portion of the interproximal tissues The buccal and lingual flaps will be elevated. For periodontal granulation tissue preservation group, the soft tissues covering the alveolar crest will be prepared. A third incision will separate the pocket epithelium from the soft tissue (granulation tissue) attached to the bone. The pocket epithelium will be removed. The root surfaces will be carefully scaled and planed in both groups. Ethylenediaminetetraacetic acid (24%) will be applied to the root surfaces and removed after 2 minutes with abundant saline solution. In the experimental group, the preserved attached soft tissue and the space between it and the root surface will be irrigated with 10% polyvinylpyrrolidone-iodine. Finally, the flaps will be positioned and sutured.

SUMMARY:
The objective of this study will be to evaluate a new protocol for the surgical treatment of periodontal disease with two novelties: to make a single incision in the midline of the interproximal area to respect the vascular supply and preserve the granulation tissue with regenerative potential.

The investigators will carry out a controlled and randomized clinical trial with a control group (n=25; modified Kirkland flap) and a test group (n=25; experimental surgical protocol: incision in the mid-interproximal area of the papilla and preservation of the granulation tissue).

Clinical parameters will be taken at the time of surgery and 12 months follow-up: bleeding on probing (BoP), clinical attachment level (CAL), residual probing depth (rPD),Probing pocket depth reduction (PPDr), recession (REC), interproximal gingival recession (iGR), width of keratinized gingiva (KT), gain of supra-alveolar clinical attachment (SUPRA-AG), early wound healing index (EHI).

ELIGIBILITY:
Inclusion Criteria:

* Stage III or IV periodontitis, including all grades.
* Unresolved deep pockets (probing pocket depth [PPD] >5 mm + BoP) 4 to 6 weeks after non-surgical treatment.
* Interproximal plaque index <35% maintained during periodontal treatment and maintenance.
* Adherence to periodontal maintenance appointments.

Exclusion Criteria:

* Systemic disease contraindicating periodontal surgery.
* Teeth with incorrect endodontic treatment or restoration.
* Stage I or II periodontitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment gain (CAG) | 12 months
  Clinical attachment gain

SECONDARY OUTCOMES:
rPD | 12 months
  residual probing depth
PPDr | 12 months
  Probing pocket depth reduction
iGR | 12 months
  interproximal gingival recession
Early Healing Index (EHI) | 1 week
  Five types of early healing will be recorded: EHI 1, complete closure of the incision line, with no fibrin; EHI 2-3, formation of a thin line or a fibrin clot in the incision area, respectively; EHI 4-5, incomplete closure with partial necrosis or necrosis of the incision area, respectively.
SUPRA-AG | 12 months
  Supra-alveolar attachment gain

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Odontologico Del Sureste Slp, Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A pilot prospective study on the periodontal granulation tissue preservation in surgical periodontal disease treatment — http://doi.org/10.5051/jpis.2105780289